CLINICAL TRIAL: NCT00026026
Title: Linkage and Identification of (a) Candidate Gene(s) for Tooth Disorders
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR02558-0173
Record Dates: First submitted 2001-11-06; First posted 2001-11-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Anodontia
Keywords: Human tooth agenesis
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Time Perspective: Cross-Sectional

SUMMARY:
The congenital absence of teeth, commonly referred to as hypodontia or tooth agenesis, is a common developmental anomaly of human dentition that affects approximately 20% of the population. Although new genetic and molecular approaches in humans and mice have increased our understanding of the molecules that control tooth patterning (number, position, shape and size), the precise nature of the genes involved in hypodontia in humans is poorly understood. Hence, understanding the molecular basis for missing teeth is an issue of paramount importance that is both timely and significant to the practice of dentistry. So far, only two genes have been associated with non-syndromic familial tooth agenesis: MSX1 and PAX9. Substitution mutations in the homeodomain region of MSX1 were linked to premolar agenesis while an insertion mutation in the paired box domain of PAX9 was shown to be responsible for molar oligodontia.

The long-term goals of this research are to elucidate the molecular pathology of human tooth agenesis, in particular, to evaluate whether genes other than MSX1 and PAX9 (locus heterogeneity) are involved. Alternatively, as in the case of MSX1, it will be interesting to know whether allelic variations, different mutations in these genes, are associated with tooth agenesis. We propose to study a potentially large kindred that report the developmental absence of several posterior teeth. The fundamental hypothesis to be tested states that the gene responsible for the congenital absence of molar teeth in this kindred is a critical element in the genesis of molars. The specific goals are to perform linkage analysis followed by direct sequencing of PCR products to identify the gene and to characterize the nature of the underlying defect. Identifying the underlying gene defect in this family affected by tooth agenesis will add new knowledge to our understanding of the pathogenesis of this defect and will provide the basis for future studies.

ELIGIBILITY:
* Patients affected with non-syndromic tooth agenesis and non-affected family members

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States